CLINICAL TRIAL: NCT03076463
Title: Long-term Effects of Grape Polyphenols as Modulators of Metabolic Syndrome in Humans
Brief Title: Grape Pomace Polyphenols and Cardiometabolic Risk
Acronym: GRAPOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Jara Pérez-Jiménez, PhD, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AGL2014-55102-JIN_2
Record Dates: First submitted 2017-02-26; First posted 2017-03-10 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Subjects at Cardiometabolic Risk
Keywords: Polyphenols; Metabolic syndrome; Cardiometabolic risk; Grape pomace; Postprandial glucose; Insulin resistance; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Obesity

STUDY DESIGN:
Intervention Model Description: GRAPOM: dried and milled grape pomaces. CTR: control period. All the subjects will pass the two periods: one half will do the CTRL period followed by the GRAPOM period, and the other half will do it inversely. The assignment to each order will be done randomly. Both period will be separated by a four weeks washing period.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRAPOM (Experimental): Daily consumption for 6 weeks of 10 g of dried and milled grape pomaces solved in water. Samples will be collected at the beginning and the end of this period
  Interventions: Dietary Supplement: GRAPOM
- CTR (No Intervention): Follow-up for 6 weeks without intervention. Samples will be collected at the beginning and the end of this period

INTERVENTIONS:
Dietary Supplement: GRAPOM — The whole intervention will be divided in 2 periods, control (CTR) and dried and milled grape pomace (GRAPOM). The two periods will have a duration of 6 weeks. During the CTR period, subjects will follow their normal dietary habits and samples will be collected at the beginning and at the end. No proper placebo could be found for the product, so this CTR period was chosen. During the GRAPOM period, the subjects will daily consume 8 g of the product solved in water and samples will be collected at the beginning and at the end.
  Arms: GRAPOM

SUMMARY:
The aim of this is study is to evaluate the long-term effects of grape polyphenols in the modulation of markers of metabolic syndrome. Most of the previous works about polyphenols have only considered a fraction of polyphenols, i.e., extractable polyphenols. As a consequence, an important amount of dietary polyphenols, the so-called non-extractable polyphenols are ignored. In contrast, the effect of both extractable and non-extractable polyphenols will be considered in this study. Also, studies on the long-term effect of grape polyphenol on markers of metabolic syndrome have been mostly conducted in animals, so clinical trials on this topic are needed.

DETAILED DESCRIPTION:
Fifty supposedly healthy volunteers with at least two cardiometabolic risk factors were recruited. The cardiometabolic risk factors used to select the subjects are described below.

The whole intervention will be divided in 2 periods, control (CTR) and dried and milled grape pomace (GRAPOM). The two periods will have a duration of 6 weeks. During the CTR period, subjects will follow their normal dietary habits and samples will be collected at the beginning and at the end. No proper placebo could be found for the product, so this CTR period was chosen. During the GRAPOM period, the subjects will daily consume 8 g of the product solved in water and samples will be collected at the beginning and at the end.

ELIGIBILITY:
Inclusion Criteria:

At least two of the following requirements:

* BMI ≥ 25 kg/m2.
* Fasting glucose values ≥ 100 mg/dL.
* Triglycerides ≥ 150 mg/dL.
* HDL-cholesterol: ≤ 50 mg/dL women, ≤ 40 mg/dL men.
* Blood pressure: systolic ≥ 130 mm Hg or diastolic ≥ 85 mm Hg.

Exclusion Criteria:

* Subjects with a pharmaceutical treatment set to modify blood pressure, lipid profile or glucose.
* Volunteers participating in other studies or weight loss plans.
* Pregnant or breastfeeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Fasting insulin | Up to three months
  Changes of blood insulin fasting levels as result of long-term supplementation with grape pomace (GRAPOM).
Fasting glucose | Up to three months
  Changes of blood glucose fasting levels as result of long-term supplementation with grape pomace (GRAPOM).

SECONDARY OUTCOMES:
Postprandial glucose | Up to four months
  Changes of blood glucose response after an oral glucose load as result of long-term supplementation with grape pomace (GRAPOM).
Postprandial insulin | Up to four months
  Changes of blood insulin response after an oral glucose load as result of long-term supplementation with grape pomace (GRAPOM).
Blood pressure | Up to four months
  Changes of blood pressure as result of long-term supplementation with grape pomace (GRAPOM).
Blood cholesterol (total, HDL, LDL) | Up to four months
  Changes of blood cholesterol (total, HDL, LDL) as result of long-term supplementation with grape pomace (GRAPOM).
Blood triglycerides | Up to four months
  Changes of blood triglycerides as result of long-term supplementation with grape pomace (GRAPOM).
Blood C reactive protein | Up to five months
  Changes of blood C reactive protein as result of long-term supplementation with grape pomace (GRAPOM).
Blood fibrinogen | Up to five months
  Changes of blood fibrinogen as result of long-term supplementation with grape pomace (GRAPOM).
Blood uric acid | Up to five months
  Changes of blood uric acid as result of long-term supplementation with grape pomace (GRAPOM).
Iron metabolism | Up to six months
  Changes of blood markers of iron metabolism as result of long-term supplementation with grape pomace (GRAPOM).
Blood polyphenols | Up to six months
  Changes of blood polyphenols as result of long-term supplementation with grape pomace (GRAPOM).
Urine uric acid | Up to six months
  Changes of urine uric acid as result of long-term supplementation with grape pomace (GRAPOM).
Urine polyphenols | Up to seen months
  Changes of urine polyphenols as result of long-term supplementation with grape pomace (GRAPOM).
Body weight | Up to three months
  Changes of body weight (measured at a body-impedance equipment) as result of long-term supplementation with grape pomace (GRAPOM).
Body fat | Up to seven months
  Changes of body fat as result of long-term supplementation with grape pomace (GRAPOM).
miRNA expression | Up to eight months
  Changes of blood expression of selected miRNA as result of long-term supplementation with grape pomace (GRAPOM).
Profile of fecal microbiota | Up to nine months
  Changes of fecal microbiota as result of long-term supplementation with grape pomace (GRAPOM).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food Science, Technology and Nutrition (ICTAN-CSIC), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No